CLINICAL TRIAL: NCT00173316
Title: The Role of Vascular Endothelial Growth Factor-C (VEGF-C) and Its Receptors Induced Lymphangiogenesis on the Carcinogenesis of Oral Cancers and Premalignant Lesions
Brief Title: Expression of VEGF-C and VEGF-CR in Oral Cancers and Premalignant Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700614
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-08

CONDITIONS: Oral Cancer
Keywords: vascular endothelial growth factor-C; VEGF-CR; lymphangiogenesis; host inflammatory responses; oral carcinogenesis; oral cancers; oral premalignant lesions
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The role of vascular endothelial growth factor-C (VEGF-C) and its receptors induced lymphangiogenesis and host inflammatory responses on the carcinogenesis of oral cancers and premalignant lesions

DETAILED DESCRIPTION:
The role of vascular endothelial growth factor-C (VEGF-C) and its receptors induced lymphangiogenesis and host inflammatory responses on the carcinogenesis of oral cancers and premalignant lesions

ELIGIBILITY:
Inclusion Criteria:

* oral cancer and oral precancer specimens

Exclusion Criteria:

* other diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-08; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Pin Chiang, DMSc, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan university, Taipei, Taiwan